CLINICAL TRIAL: NCT07132671
Title: MRI-guided Brachytherapy + Salvage SBRT Program for Patients With Prostate Bed Relapses After Radical Prostatectomy
Brief Title: MRI-guided Brachytherapy and Salvage SBRT Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.224
Record Dates: First submitted 2025-06-17; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: Prostate Cancer; Prostate Bed Relapse; Brachytherapy; MR-Guided SBRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-guided Brachytherapy and Salvage SBRT Program (Experimental): Brachytherapy and MR-guided SBRT
  Interventions: Radiation: Brachytherapy and MR-Guided SBRT

INTERVENTIONS:
Radiation: Brachytherapy and MR-Guided SBRT — HDR Brachytherapy followed by MR-guided SBRT

SUMMARY:
Brachytherapy followed by MRI-guided irradiation has the potential to improve treatment results in patients with local relapses after radical prostatectomy

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if the use of brachytherapy followed by MRI-guided irradiation increases the rates of tumor control and decreases the rates of adverse events in patients with tumor bed relapses after radical prostatectomy

ELIGIBILITY:
Patients with increasing PSA after RP and clinical evidence of PET PSMA/Choline+ and RMN+ isolated prostatic bed relapse (IPBR) that is implantable via transperineal route . The IPBR should be visible on TRUS imaging to allow proper implant placement.

1. Pathological confirmation is advised in all cases but it is not mandatory .
2. Patients with any of the following were not considered eligible:

   1. Distance < 5mm from the edge of the IPBR to any of the defined OARs (UV anastomosis, rectal wall, bladder wall, external urinary sphincter)
   2. Distant Metastases
   3. Isolated nodal relapses
   4. Prior Irradiation to the IPBR area
   5. Multicentric IPBRs
   6. Life expectancy of less than 5 years or inability to tolerate and comply with an HDR procedure
3. No prior radiation therapy to the target areas;
4. Karnofsky performance status > 70 with medical condition not contraindicating treatment with radical intent including maximal TURBT and concomitant chemotherapy;
5. WBC equal or greater than 3500 mm3; platelet count equal or greater than 135000 mm3; hemoglobin equal or greater than 10 gr/L; BUN equal or less than 20; serum creatinine equal or less than 2.0.
6. Ability to undergo MRI scanning.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical control | 5-year
  To achieve 5-year biochemical control rate in 85% of the patients.
Adverse Events | 5-year
  To decrease urinary grade 3 or greater toxicity below 3% and rectal grade 3 or greater toxicity below 1%.

SECONDARY OUTCOMES:
QOL | From enrollment to extended follow-up at 5 years with QOL assessment at 3, 6, 12 months after treatment and yearly thereafter
  Determination of QOL with the EORTC QLQ-PR25

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Marta Gimeno-Morales, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 1st, 2025 - June 30th, 2030
Access Criteria: On request